CLINICAL TRIAL: NCT03876704
Title: Effects of Fat-soluble Vitamins Supplementation in Early Life on Common Complications and Neural Development in Very Low Birth Weight Infants
Brief Title: Effects of Fat-soluble Vitamins Supplementation on Common Complications and Neural Development in Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xi'an Gaoxin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018MSZC-04
Record Dates: First submitted 2019-03-03; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Vitamin A Deficiency; Vitamin D Deficiency; Vitamin E Deficiency; Very Low Birth Weight Infants; Bronchopulmonary Dysplasia; Anemia; Sepsis
MeSH Terms: conditions — Vitamin A Deficiency; Vitamin D Deficiency; Vitamin E Deficiency; Bronchopulmonary Dysplasia; Anemia; Sepsis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose of fat-soluble vitamins (Experimental): Fat-soluble vitamins is administered 0.5 piece/kg (equals to 1150 U/kg vitamin A，200 U/kg vitamin D, 3.2 U/kg vitamin E) intravenously every day until the baby achieve full enteral feeding (120 ml/kg), starting with the first dose within 24 hours after birth.
  Interventions: Drug: High dose of fat-Soluble Vitamin
- Conventional dose of fat-soluble vitamins (Active Comparator): Fat-soluble vitamins is administered 0.1 piece/kg (equals to 230 U/kg vitamin A，40 U/kg vitamin D, 0.64 U/kg vitamin E) intravenously every day until the baby achieve full enteral feeding (120 ml/kg), starting with the first dose within 24 hours after birth.
  Interventions: Drug: Conventional dose of fat-Soluble Vitamin

INTERVENTIONS:
Drug: High dose of fat-Soluble Vitamin — Supplementation of 5 times current dose of fat-soluble vitamins by intravenous perfusion
  Arms: High dose of fat-soluble vitamins
Drug: Conventional dose of fat-Soluble Vitamin — Supplementation of the current dose of fat-soluble vitamins by intravenous perfusion
  Arms: Conventional dose of fat-soluble vitamins

SUMMARY:
Vitamins A, D, and E play important roles in humans, such as vision function, immune function, bone metabolism, cell growth and differentiation and oxidation resistance. Deficiencies in these vitamins will result in a high prevalence of cardiovascular disease, infection, bone diseases, etc. Preterm infants, especially very low birth weight infants, are at risk of vitamin deficiency. Intravenous perfusion is the most common and widely used method to supply vitamins for the specific population in early life. However, the current dose of vitamin supplied by intravenous perfusion whether can meet the need of growth and development is not sure and the appropriate dose for preterm infants is still uncertain. The purpose of this study is to investigate whether current dose of fat-soluble vitamin supplementation is enough for very low birth weight infants, the safety of high dose of fat-soluble vitamin supplementation, and compare the differences of prevalence of common complications, such as bronchopulmonary dysplasia, patent ductus arteriosus, sepsis, anemia, and neural development between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the neonatal intensive care unit (NICU) within 24 hours after birth
* gestational age younger than 34 weeks
* birth weight less than 1500 gram
* informed consent was obtained from the infants' parents or guardians

Exclusion Criteria:

* congenital malformation
* chromosomal disease, genetic metabolic diseases
* the infants or his/mother has abnormal thyroid function or parathyroid gland function
* neonatal necrotizing enterocolitis, diarrhea
* intracranial hemorrhage of 3 degrees or above
* pulmonary hemorrhage
* liver enzymes elevated by more than 2 times, cholestasis
* death or discharge against medical advice
* refuse to take part in the study

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin levels | within 72 hours after birth, 4~6 weeks old
  Change from baseline level of vitamin A, vitamin D, and vitamin E at 4~6 weeks

SECONDARY OUTCOMES:
Complications | corrected age of 36 weeks
  The prevalence of bronchopulmonary dysplasia, patent ductus arteriosus, sepsis, anemia, intracranial hemorrhage, extrauterine growth retardation, etc.
Neural development | corrected age of 40 weeks
  White matter disease of the preterm infant, was semiquantitatively assessed from MRI at term-equivalent age based on an established scoring method.
Gene polymorphism in vitamin deficiency preterm infants | within 72 hours after birth, 4~6 weeks old
  Association of rs4588 polymorphism in vitamin D receptor gene and rs10766197 polymorphism in the cytochrome P450 family 2 subfamily R member 1 gene with baseline level of vitamin D and change in vitamin D level after 4~6 weeks' supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Liu, Study Director — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kositamongkol S, Suthutvoravut U, Chongviriyaphan N, Feungpean B, Nuntnarumit P. Vitamin A and E status in very low birth weight infants. J Perinatol. 2011 Jul;31(7):471-6. doi: 10.1038/jp.2010.155. Epub 2011 Jan 13. PMID 21233795
- [Background] Mactier H, Mokaya MM, Farrell L, Edwards CA. Vitamin A provision for preterm infants: are we meeting current guidelines? Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F286-9. doi: 10.1136/adc.2010.190017. Epub 2011 Jan 17. PMID 21242240
- [Background] Jilani T, Iqbal MP. Vitamin E deficiency in South Asian population and the therapeutic use of alpha-tocopherol (Vitamin E) for correction of anemia. Pak J Med Sci. 2018 Nov-Dec;34(6):1571-1575. doi: 10.12669/pjms.346.15880. PMID 30559825
- [Background] Cho SY, Park HK, Lee HJ. Efficacy and safety of early supplementation with 800 IU of vitamin D in very preterm infants followed by underlying levels of vitamin D at birth. Ital J Pediatr. 2017 May 4;43(1):45. doi: 10.1186/s13052-017-0361-0. PMID 28472980
- [Result] Fares S, Sethom MM, Khouaja-Mokrani C, Jabnoun S, Feki M, Kaabachi N. VitaminA, E, and D deficiencies in tunisian very low birth weight neonates: prevalence and risk factors. Pediatr Neonatol. 2014 Jun;55(3):196-201. doi: 10.1016/j.pedneo.2013.09.006. Epub 2013 Nov 26. PMID 24289974